CLINICAL TRIAL: NCT03908697
Title: Comparison of Two Hormonal Fertility Monitors for Use in Natural Family Planning
Brief Title: Quantum Natural Family Planning Pilot
Acronym: QNFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quanovate Tech Inc. (Industry)
Responsible Party: Principal Investigator, Thomas Bouchard, MD, Clinical Lecturer, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HREBA.CTC-19-0046
Record Dates: First submitted 2019-04-02; First posted 2019-04-09 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Intervention Model Description: Prospective cohort analysis of three menstrual cycles of hormone data, comparing two fertility monitors that analyze urine hormones. Satisfaction and ease of use will be assessed using surveys. Individual data will be anonymized.
Masking Description: Anonymized demographic data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single cohort (Experimental): All 20 participants will use ClearBlue and Mira monitors on first morning urine
  Interventions: Device: Mira monitor comparison to ClearBlue monitor

INTERVENTIONS:
Device: Mira monitor comparison to ClearBlue monitor — Testing first morning urine with hormone test sticks at home

SUMMARY:
•The Pilot study will involve current Marquette Method users who own and use a ClearBlue Fertility monitor and who will be asked to simultaneously use the Mira monitor for the sake of comparing the two devices to monitor the menstrual cycle.

DETAILED DESCRIPTION:
* The Mira fertility monitoring system (www.miracare.com) is a new home-use hormone tracking device with the ability to quantitatively measure reproductive hormones in the urine but is also synced to a smart phone App that provides a graphic representation of the hormonal levels throughout a menstrual cycle.
* The Mira monitor will be compared to the ClearBlue Fertility Monitor for its ease of use, satisfaction, and accuracy.
* The Mira hormonal monitor and App system has not been tested for its use in Natural Family Planning (NFP).
* The Pilot study will involve current Marquette Method users who own and use a ClearBlue Fertility monitor and who will be asked to simultaneously use the Mira monitor for the sake of comparing the two devices.
* Female participants invited to participate will need to meet the following criteria:
* Age 18 to 42 years
* Menstrual cycle ranging between 21-42 days
* At least 3 cycles after cessation of breastfeeding
* Not currently on medications that affect ovulation and 3 months prior
* Not currently pregnant or breastfeeding
* No known fertility problems
* Not planning on achieving pregnancy during the 3 menstrual cycles of the study

ELIGIBILITY:
Inclusion Criteria:

* • Menstrual cycle ranging between 21-42 days

  * At least 3 cycles after cessation of breastfeeding

Exclusion Criteria:

* • Not currently on medications that affect ovulation and 3 months prior

  * Not currently pregnant or breastfeeding
  * No known fertility problems
  * Not planning on achieving pregnancy during the 3 menstrual cycles of the study

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Day of the estimated beginning of the fertile phase of the menstrual cycle: | 3 months
  First day of the estimated fertile phase as measured by Clearblue Fertility Monitor First day of the estimated fertile phase as measured by the MIRA Fertility Monitor
Day of the estimated peak of the fertile phase of the menstrual cycle: | 3 months
  Peak day of the estimated fertile phase as measured by the Clearblue Fertility Monitor Peak day of the estimated fertile phase as measured by the MIRA Fertility Monitor
Day of the estimated end of the fertile phase of the menstrual cycle: | 3 months
  Last day of the estimated fertile phase as measured by the Clearblue Fertility Monitor Last day of the estimated fertile phase as measured by the MIRA Fertility Monitor

SECONDARY OUTCOMES:
Satisfaction and Ease of Use of a Electronic Fertility Monitor: | 3 months
  Measured by the modified 8 item Severy Satisfaction Scale
  Total score rages from 8 - 24 with 24 being the highest satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Deer Valley family Medicine Clinic, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouchard TP, Fehring RJ, Schneider MM. Achieving Pregnancy Using Primary Care Interventions to Identify the Fertile Window. Front Med (Lausanne). 2018 Jan 9;4:250. doi: 10.3389/fmed.2017.00250. eCollection 2017. PMID 29376054
- [Background] Ecochard R, Bouchard T, Leiva R, Abdulla S, Dupuis O, Duterque O, Garmier Billard M, Boehringer H, Genolini C. Characterization of hormonal profiles during the luteal phase in regularly menstruating women. Fertil Steril. 2017 Jul;108(1):175-182.e1. doi: 10.1016/j.fertnstert.2017.05.012. Epub 2017 Jun 1. PMID 28579410
- [Background] Leiva RA, Bouchard TP, Abdullah SH, Ecochard R. Urinary Luteinizing Hormone Tests: Which Concentration Threshold Best Predicts Ovulation? Front Public Health. 2017 Nov 28;5:320. doi: 10.3389/fpubh.2017.00320. eCollection 2017. PMID 29234665
- [Background] Direito A, Bailly S, Mariani A, Ecochard R. Relationships between the luteinizing hormone surge and other characteristics of the menstrual cycle in normally ovulating women. Fertil Steril. 2013 Jan;99(1):279-285.e3. doi: 10.1016/j.fertnstert.2012.08.047. Epub 2012 Sep 19. PMID 22999798
- [Background] Severy LJ, Robinson J, Findley-Klein C, McNulty J. Acceptability of a home monitor used to aid in conception: psychosocial factors and couple dynamics. Contraception. 2006 Jan;73(1):65-71. doi: 10.1016/j.contraception.2005.07.008. Epub 2005 Sep 19. PMID 16371298
- See also: Official product website — https://www.miracare.com